CLINICAL TRIAL: NCT01262287
Title: Placebo Controlled Pilot Study of Dutasteride for the Reduction of Alcohol Use in Male Drinkers
Brief Title: Dutasteride for the Reduction of Alcohol Use in Male Drinkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jonathan Covault, Professor of Psychiatry, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-036-2; P60AA003510 (NIH)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Alcoholism; Alcohol Abuse; Alcohol Dependence
Keywords: Randomized Trial; Medication for Heavy Drinking; Dutasteride Treatment
MeSH Terms: conditions — Alcoholism | interventions — Dutasteride; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dutasteride (Experimental): dutasteride (1 mg oral daily dose) for 8-week treatment period
  Interventions: Drug: Dutasteride
- Placebo (Placebo Comparator): placebo daily for 8-week treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride — dutasteride 4 mg loading dose followed by 1 mg daily for 8-week treatment period
  Other Names: Avodart
  Arms: dutasteride
Drug: Placebo — placebo capsules in same number as active drug, daily for 8-week treatment period
  Other Names: Lactose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether dutasteride is safe and effective for reducing alcohol use in male drinkers who want to stop or reduce their drinking. The investigators hypothesize that at a dosage of 1mg/day, dutasteride will be well tolerated and that, compared to placebo treatment, dutasteride will result in a greater reduction in the amount of alcohol consumed per week. The study sample size is of a pilot scale and is designed to provide additional support for the study hypothesis and provide an estimate of likely effect sizes in order to design a more definitive study.

ELIGIBILITY:
Inclusion Criteria:

* Male outpatients age 18 to 65 years
* Have an average weekly ethanol consumption of >24 standard drinks
* Be able to read English at the 8th grade or higher level and show no evidence of significant cognitive impairment
* Be willing to nominate an individual who will know the patient's whereabouts in order to facilitate follow up during the study
* Be willing to provide signed, informed consent to participate in the study (including a willingness to reduce drinking to non-hazardous levels)

Exclusion Criteria:

* Have a current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation
* Have a serious psychiatric illness (e.g., schizophrenia, bipolar disorder, severe or psychotic major depression, organic mood or mental disorders, current eating disorder symptoms, or substantial suicide or violence risk) on the basis of history or psychiatric examination
* Have a current diagnosis of drug dependence (other than nicotine or alcohol dependence)
* Have a current diagnosis of alcohol dependence who on clinical examination by a physician, are deemed to be too severely alcohol dependent to permit them to participate in a placebo-controlled pilot study
* Have a history of hypersensitivity to dutasteride
* Current or past 4 month use of finasteride (Propecia), dutasteride (Avodart) or testosterone
* Are currently taking psychotropics other than a single antidepressant with stable dose for at least 4 weeks or a non-benzodiazepine sleep medication
* Are considered by the investigators to be an unsuitable candidate for receipt of an investigational drug

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Covault, MD, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 subjects excluded during screening due to medical or laboratory exclusion (n=3) or current drug dependence (n=1); 4 subjects lost interest in participation following screening and prior to randomization to treatment arm resulting in 37 subjects available for randomization to treatment arm
Period: Overall Study
Arm/Group | Dutasteride | Placebo
Started | 20 | 19
Completed | 18 | 18
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dutasteride | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 17 | 36
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.95 (10.21) | 54.95 (7.44) | 52.90 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change Number of Standard Drinks Per Week.
Description: Change in Average Standard Drinks (14 gr ethanol) per week: last 2 weeks of treatment (wk 7-8) minus baseline average drinking average from baseline 90 day drinking history
Time Frame: Baseline (average weekly drinking for 90 day period prior to screening) vs. End Point (average weekly drinking weeks 7 and 8 of treatment)
Measure: Mean (Standard Error); unit: standard drinks per week
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 18 | 18
standard drinks per week | -26.2 (4.6) | -25.5 (4.1)
Statistical Analysis 1: Comparison: Dutasteride vs Placebo; Test type: Superiority or Other; p = 0.9, t-test, 2 sided

2. Secondary Outcome: Change in Standard Drinks Per Week - Moderation by Genetic Variation
Description: Moderation of primary outcome measure [change in standard drinks per week from baseline to end point (average weeks 7 and 8 of treatment)] by genetic variation rs12529 in neuroactive steroid biosynthetic enzyme gene AKR1C (AKR1C3*2 C-allele associated with alcohol use disorder)
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: standard drinks per week
Groups:
- AKR1C3*2 C/C Genotype + Dutasteride: AKR1C3*2 C/C genotype subjects in dutasteride arm (1 mg daily for 8 wks)
- AKR1C3*2 C/C Genotype + Placebo: AKR1C3*2 C/C genotype subjects in placebo arm
  placebo: placebo capsules in same number as active drug, daily for 8-week treatment period
- AKR1C3*2 G-carriers + Dutasteride: AKR1C3*2 G-carriers in dutasteride arm (1 mg/day x 8 wks)
- AKR1C3*2 G-carriers + Placebo: AKR1C3*2 G-carriers in placebo arm
Arm/Group | AKR1C3*2 C/C Genotype + Dutasteride | AKR1C3*2 C/C Genotype + Placebo | AKR1C3*2 G-carriers + Dutasteride | AKR1C3*2 G-carriers + Placebo
Number analyzed (Participants) | 8 | 5 | 10 | 13
standard drinks per week | -32.4 (5.4) | -31.2 (13.9) | 21.8 (6.9) | -22.3 (3.3)
Statistical Analysis 1: Comparison: AKR1C3*2 C/C Genotype + Dutasteride vs AKR1C3*2 C/C Genotype + Placebo; Test type: Superiority or Other; p = 0.9, t-test, 2 sided
Statistical Analysis 2: Comparison: AKR1C3*2 G-carriers + Dutasteride vs AKR1C3*2 G-carriers + Placebo; Test type: Superiority or Other; p = 0.9, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Dutasteride | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 11/20 | 9/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dutasteride (N=20) | Placebo (N=19)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Tiredness (General disorders) | 2 (2) | 2 (4)
Stomach discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
change in sleep (General disorders) | 3 (14) | 3 (6)
lightheadness/dizziness (General disorders) | 1 (4) | 1 (3)
Muscle or joint ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (6)
Reduced libido (Reproductive system and breast disorders) | 2 (6) | 3 (9)
Impotence (Reproductive system and breast disorders) | 0 (0) | 1 (5)
gynecomastia (Reproductive system and breast disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
28% of participants were abstinent for the entire 8-week medication treatment period which reduced ability to detect the hypothesized treatment effects of dutasteride related to alcohol's acute effects on neuroactive steroid production.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No